CLINICAL TRIAL: NCT03747874
Title: Prevalence of Obstructive Sleep Apnea Syndrome in Patients With a History of Sudden Sensorineural Hearing Loss
Brief Title: OSA and Sudden Sensorineural Hearing Loss
Acronym: SAS-SB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SAS-SB
Record Dates: First submitted 2018-11-17; First posted 2018-11-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Obstructive Sleep Apnea; Sudden Hearing Loss
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hearing Loss, Sudden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- past medical history of sudden hearing loss (Other): sleep examination and ventilatory polygraphy device for 1 night
  Interventions: Diagnostic Test: ventilatory polygraphy

INTERVENTIONS:
Diagnostic Test: ventilatory polygraphy — we put a ventilatory polygraphy device on the patient in the evening, they come back home to sleep while the device is recording ventilatory parameters and they come back the morrow to give the device back

SUMMARY:
This study studies the prevalence between obstructive sleep apnea syndrome and sensorineural hearing loss. We recruit patients who have been treated for sudden sensorineural hearing loss in Poitiers' University Hospital between 2010 et 2017, and we detect if they have OSA with a ventilatory polygraphy.

ELIGIBILITY:
Inclusion Criteria:

* past medical history of sudden hearing loss between 2010 and 2017
* no contraindication to a non supervised sleeping monitoring

Exclusion Criteria:

* past medical history of fluctuant hearing loss or pre-existant significative hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Study of the prevalence of OSA on patient with a history of sudden hearing loss | 1 night

CONTACTS AND LOCATIONS:
Locations (1):
- Dufour Xavier, Poitiers, France

IPD SHARING:
Plan to Share IPD: No